CLINICAL TRIAL: NCT00359762
Title: Long Term Treatment With Exenatide Versus Glimepiride in Patients With Type 2 Diabetes Pretreated With Metformin (EUREXA: European Exenatide Study)
Brief Title: Exenatide Versus Glimepiride in Patients With Type 2 Diabetes
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: AstraZeneca (Industry)
Collaborators: Eli Lilly and Company (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: H8O-EW-GWBE
Record Dates: First submitted 2006-07-31; First posted 2006-08-02 (Estimated); Results first posted 2013-03-14 (Estimated); Last update posted 2015-09-15 (Estimated); Status verified 2015-08

CONDITIONS: Type 2 Diabetes Mellitus
Keywords: exenatide; diabetes; Amylin; Lilly; glimepiride
MeSH Terms: conditions — Diabetes Mellitus, Type 2; Diabetes Mellitus | interventions — Exenatide; glimepiride

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Exenatide (Experimental)
  Interventions: Drug: exenatide
- Glimepiride (Active Comparator)
  Interventions: Drug: glimepiride

INTERVENTIONS:
Drug: exenatide — subcutaneous injection (5mcg or 10mcg), twice a day
  Other Names: Byetta
  Arms: Exenatide
Drug: glimepiride — oral tablet (titrated to maximally tolerated dose), once daily
  Other Names: Amaryl
  Arms: Glimepiride

SUMMARY:
This study assesses the effects of twice-daily subcutaneous injection exenatide versus treatment with sulfonylurea (glimepiride) on long-term glycemic control and beta-cell function.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosed with type 2 diabetes mellitus.
* Treated with diet and exercise and a stable, maximally tolerated dose of metformin for at least 3 months prior to screening.
* HbA1c >=6.5% and <=9.0%.
* Body Mass Index (BMI) >=25 kg/m^2 and <40 kg/m^2.

Exclusion Criteria:

* Participated in an interventional medical, surgical, or pharmaceutical study within 30 days prior to screening.
* Characteristics contraindicating metformin or glimepiride use.
* Receiving drugs that directly affect gastrointestinal motility.
* Receiving chronic (lasting longer than 2 weeks) systemic glucocorticoid therapy.
* Have used any prescription drug to promote weight loss within 3 months prior to screening.
* Treated for longer than 2 weeks with any of the following medications within 3 months prior to screening: *insulin; *thiazolidinediones; *alpha-glucosidase inhibitors; *sulfonylurea; *meglitinides

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1029 (Actual)
Dates: Start 2006-09; Primary Completion 2011-03 (Actual); Study Completion 2011-03 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: James Malone, MD, Study Director — Eli Lilly and Company
Locations (114):
- Austria (4):
  - Research Site, Graz
  - Research Site, Innsbruck
  - Research Site, Salzburg
  - Research Site, Vienna
- Czechia (7):
  - Research Site, Beroun
  - Research Site, České Budějovice
  - Research Site, Hradec Králové
  - Research Site, Liberec
  - Research Site, Písek
  - Research Site, Prague
  - Research Site, Třebíč
- Finland (4):
  - Research Site, Helsinki
  - Research Site, Kuopio
  - Research Site, Pori
  - Research Site, Vaasa
- France (17):
  - Research Site, Alençon
  - Research Site, Bois-Guillaume
  - Research Site, Bourg-des-Comptes
  - Research Site, Broglie
  - Research Site, Bron
  - Research Site, Fléville-devant-Nancy
  - Research Site, Le Creusot
  - Research Site, Le Mans
  - Research Site, Loudun
  - Research Site, Montigny-lès-Metz
  - Research Site, Nevers
  - Research Site, Strasbourg
  - Research Site, Thouars
  - Research Site, Tours
  - Research Site, Valréas
  - Research Site, Vénissieux
  - Research Site, Vihiers
- Germany (19):
  - Research Site, Altona
  - Research Site, Aschaffenburg
  - Research Site, Bad Staffelstein
  - Research Site, Dresden
  - Research Site, Eisenach
  - Research Site, Essen
  - Research Site, Essen Schonnebeck
  - Research Site, Falkensee
  - Research Site, Fulda
  - Research Site, Hamburg
  - Research Site, Hamburg-Ottmarschen
  - Research Site, Heidelberg
  - Research Site, Leipzig
  - Research Site, Münster
  - Research Site, Saarbrücken
  - Research Site, Saint Ingbert
  - Research Site, Schenklengsfeld
  - Research Site, Schkeuditz
  - Research Site, Witten
- Hungary (5):
  - Research Site, Budapest
  - Research Site, Gyula
  - Research Site, Kecskemét
  - Research Site, Veszprém
  - Research Site, Zalaegerszeg
- Ireland (3):
  - Research Site, County Galway
  - Research Site, County Waterford
  - Research Site, Dublin
- Israel (4):
  - Research Site, Haifa
  - Research Site, Holon
  - Research Site, Jerusalem
  - Research Site, Tel Litwinsky
- Italy (23):
  - Research Site, Ancona
  - Research Site, Arenzano
  - Research Site, Atri
  - Research Site, Bergamo
  - Research Site, Catanzaro
  - Research Site, Florence
  - Research Site, Foggia
  - Research Site, Forlì
  - Research Site, Genova
  - Research Site, Grosseto
  - Research Site, Milan
  - Research Site, Monserrato (Cagliari)
  - Research Site, Napoli
  - Research Site, Palermo
  - Research Site, Perugia
  - Research Site, Pescara
  - Research Site, Pisa
  - Research Site, Ravenna
  - Research Site, Roma
  - Research Site, San Benedetto del Tronto
  - Research Site, Siena
  - Research Site, Treviso
  - Research Site, Verona
- Mexico (4):
  - Research Site, Celaya, Guanajuato
  - Research Site, Pachuca, Hidalgo
  - Research Site, Mexico City, Mexico City
  - Research Site, Monterrey, Nuevo León
- Poland (6):
  - Research Site, Bialystok
  - Research Site, Bydgoszcz
  - Research Site, Lublin
  - Research Site, Szczecin
  - Research Site, Warsaw
  - Research Site, Wroclaw
- Spain (2):
  - Research Site, Barcelona
  - Research Site, Madrid
- Switzerland (4):
  - Research Site, Fribourg
  - Research Site, Geneva
  - Research Site, Lausanne
  - Research Site, Lucerne
- United Kingdom (12):
  - Research Site, Bath
  - Research Site, Belfast
  - Research Site, Brandford on Avon
  - Research Site, County Antrim
  - Research Site, Downpatrick
  - Research Site, Frome
  - Research Site, Midsomer Norton
  - Research Site, Omagh
  - Research Site, Penzance
  - Research Site, Plymouth
  - Research Site, Southdown
  - Research Site, Wiltshire

REFERENCES:
- [Derived] Simo R, Guerci B, Schernthaner G, Gallwitz B, Rosas-Guzman J, Dotta F, Festa A, Zhou M, Kiljanski J. Long-term changes in cardiovascular risk markers during administration of exenatide twice daily or glimepiride: results from the European exenatide study. Cardiovasc Diabetol. 2015 Sep 4;14:116. doi: 10.1186/s12933-015-0279-z. PMID 26338040
- [Derived] Schernthaner G, Rosas-Guzman J, Dotta F, Guerci B, Simo R, Festa A, Kiljanski J, Zhou M, Gallwitz B. Treatment escalation options for patients with type 2 diabetes after failure of exenatide twice daily or glimepiride added to metformin: results from the prospective European Exenatide (EUREXA) study. Diabetes Obes Metab. 2015 Jul;17(7):689-98. doi: 10.1111/dom.12471. Epub 2015 May 8. PMID 25846577
- [Derived] Gallwitz B, Guzman J, Dotta F, Guerci B, Simo R, Basson BR, Festa A, Kiljanski J, Sapin H, Trautmann M, Schernthaner G. Exenatide twice daily versus glimepiride for prevention of glycaemic deterioration in patients with type 2 diabetes with metformin failure (EUREXA): an open-label, randomised controlled trial. Lancet. 2012 Jun 16;379(9833):2270-8. doi: 10.1016/S0140-6736(12)60479-6. Epub 2012 Jun 9. PMID 22683137

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: Patients meeting defined failure of HbA1c control (primary endpoint) in Study Period II were eligible for entry to Study Period III
Groups:
- Period II, Glim + Met: Glimepiride one 1 mg tablet daily with subsequent titration every 4 weeks to maximally-tolerated dose for the remainder of Period II and daily oral Metformin
- Period III, Exen + Met + Glim - Randomized: Glimepiride once daily, started at 1 mg dose and titrated up to maintenance doses, was added to Exenatide 10 mcg twice daily subcutaneously injected and daily oral Metformin in Period III
- Period III, Exen + Met + Pio or Rosi - Randomized: Oral Rosiglitazone or Pioglitazone once or twice daily, started 15 mg per day, was added to Exenatide 10 mcg twice daily subcutaneously injected and daily oral Metformin in Period III
- Period III, Glim + Met + Exen - Not Randomized: Exenatide 10 mcg twice daily subcutaneously injected (5 mcg exenatide per dose for the first 4 weeks followed by 10 mcg exenatide per dose for the remainder of period III) was added to oral Glimepiride once daily and daily oral Metformin in Period III
- Period II, Exen + Met: Exenatide 10 mcg twice daily subcutaneously injected (5 mcg exenatide per dose for first 4 weeks followed by 10 mcg exenatide per dose for the remainder of period II) and daily oral Metformin
Period: Period II
Arm/Group | Period II, Glim + Met | Period III, Exen + Met + Glim - Randomized | Period III, Exen + Met + Pio or Rosi - Randomized | Period III, Glim + Met + Exen - Not Randomized | Period II, Exen + Met
Started | 514 | 0 | 0 | 0 | 515
Intent to Treat (ITT) Safety Population | 508 | 0 | 0 | 0 | 511
ITT Efficacy Population | 487 | 0 | 0 | 0 | 490
Met Primary Endpoint | 262 | 0 | 0 | 0 | 203
Without Treatment Failure | 124 | 0 | 0 | 0 | 138
Completed | 386 | 0 | 0 | 0 | 341
Not Completed | 128 | 0 | 0 | 0 | 174
Not completed — Adverse Event | 17 | 0 | 0 | 0 | 49
Not completed — Protocol Violation | 18 | 0 | 0 | 0 | 11
Not completed — Physician Decision | 17 | 0 | 0 | 0 | 23
Not completed — Death | 2 | 0 | 0 | 0 | 4
Not completed — Lack of Efficacy | 11 | 0 | 0 | 0 | 8
Not completed — Lost to follow up | 5 | 0 | 0 | 0 | 5
Not completed — Entry Criteria Not Met | 8 | 0 | 0 | 0 | 4
Not completed — Subject Decision | 50 | 0 | 0 | 0 | 70
Period: Period III
Arm/Group | Period II, Glim + Met | Period III, Exen + Met + Glim - Randomized | Period III, Exen + Met + Pio or Rosi - Randomized | Period III, Glim + Met + Exen - Not Randomized | Period II, Exen + Met
Started | 0 | 77 | 77 | 166 | 0
Extension ITT Safety Population | 0 | 74 | 76 | 166 | 0
Extension ITT Efficacy Population | 0 | 73 | 75 | 164 | 0
Completed | 0 | 48 | 47 | 101 | 0
Not Completed | 0 | 29 | 30 | 65 | 0
Not completed — Protocol Violation | 0 | 5 | 3 | 8 | 0
Not completed — Adverse Event | 0 | 3 | 4 | 10 | 0
Not completed — Physician Decision | 0 | 5 | 9 | 15 | 0
Not completed — Lack of Efficacy | 0 | 7 | 5 | 9 | 0
Not completed — Lost to follow up | 0 | 1 | 1 | 2 | 0
Not completed — Entry Criteria Not Met | 0 | 1 | 0 | 1 | 0
Not completed — Subject Decision | 0 | 7 | 8 | 20 | 0
Period: Period I
Arm/Group | Period II, Glim + Met | Period III, Exen + Met + Glim - Randomized | Period III, Exen + Met + Pio or Rosi - Randomized | Period III, Glim + Met + Exen - Not Randomized | Period II, Exen + Met
Started | 0 | 0 | 0 | 0 | 0
Completed | 0 | 0 | 0 | 0 | 0
Not Completed | 0 | 0 | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Exen + Met: Exenatide 10 mcg twice daily subcutaneously injected (5 mcg exenatide per dose for first 4 weeks followed by 10 mcg exenatide per dose for the remainder of period II) and daily oral Metformin
- Glim + Met: Glimepiride one 1 mg tablet daily with subsequent titration every 4 weeks to maximally-tolerated dose for the remainder of Period II and daily oral Metformin
- Total: Total of all reporting groups
Arm/Group | Exen + Met | Glim + Met | Total
Number analyzed (Participants) | 490 | 487 | 977
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 388 | 389 | 777
  >=65 years | 102 | 98 | 200
Age, Continuous [Mean (Standard Deviation); unit: years] | 56.1 (10.03) | 56.8 (9.14) | 56.4 (9.60)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 218 | 235 | 453
  Male | 272 | 252 | 524
Glycosylated hemoglobin (HbA1c) [Mean (Standard Deviation); unit: percentage of total hemoglobin] | 7.4 (0.69) | 7.4 (0.71) | 7.4 (0.70)
Weight [Mean (Standard Deviation); unit: kg] | 92.8 (16.70) | 91.1 (14.78) | 92.0 (15.78)

OUTCOME MEASURES:

1. Primary Outcome: Number of Patients With Treatment Failure
Description: Treatment failure is defined as one of the following:1. HbA1c exceeding 9% at any visit after the initial 3 months of treatment (i.e., earliest at Month 6), on the maximally tolerated dose of antidiabetic agents. 2. HbA1c exceeding 7% at 2 consecutive visits 3 months apart, after the initial 6 months of treatment (i.e., earliest at Month 9), on the maximally tolerated dose of antidiabetic agents.
Time Frame: Baseline to end of Period II (up to 4.5 years)
Population: ITT Efficacy Population: Enrolled patients with a baseline and at least one post-baseline measurement of HbA1c in Study Period II (including only Study Period II); patients analyzed according to treatment as randomized.
Measure: Number; unit: number of patients
Arm/Group | Exen + Met | Glim + Met
Number analyzed (Participants) | 490 | 487
number of patients
  Number of patients with treatment failure | 203 | 262
  Number of patients censored | 287 | 225
Statistical Analysis 1: Comparison: Exen + Met vs Glim + Met; The null hypothesis (H0) and alternative hypothesis (H1) for the primary analysis (i.e., non-inferiority) are:H0: hazards of treatment for Exenatide/hazards of treatment for Glimepiride >=1.25.H1: hazards of treatment for Exenatide/hazards of treatment for Glimepiride < 1.25. With 527 patients in each arm, the study would have approximately 90% power to conclude non-inferiority of Exenatide to Glimepiride; Test type: Non-Inferiority or Equivalence — Non inferiority test was based on the upper 1-sided 97.5% CI for the hazard ratio of Exenatide/Glimepiride;the upper bound was compared to 1.25: if <1.25, the hypothesis that the risk of treatment failure with Exenatide is more than 1.25 times greater than the risk with Glimepiride is rejected.Superiority test was based on the 2-sided 95% CI for the hazard ratio. If CI excludes 1, the hypothesis that the risk of treatment failure with Exenatide is equal to that with Glimepiride is rejected; p = 0.0020, Regression, Cox; Time to treatment failure was modeled using Cox regression with treatment and baseline HbA1c as predictive terms; Hazard Ratio = 0.748, 95% CI 2-sided [0.623 to 0.899]

2. Primary Outcome: Time to Treatment Failure
Description: as for outcome 1
Time Frame: Baseline to end of Period II (up to 4.5 years)
Population: ITT Efficacy Population.
Measure: Median (95% Confidence Interval); unit: week
Arm/Group | Exen + Met | Glim + Met
Number analyzed (Participants) | 490 | 487
week | 180.0 [140.9 to NA] — Since the last observed time point, beyond which all are missing, is still within the 95% confidence interval for the median survival time, the upper bound should be no less than the last observed time point, and is unknown due to censoring. | 142.1 [118.6 to 161.1]
Statistical Analysis 1: Comparison: Exen + Met vs Glim + Met; Kaplan-Meier survival curves for time to treatment failure were compared between treatment groups using log rank test; Test type: Superiority or Other; p = 0.0315, Log Rank

3. Secondary Outcome: Homeostasis Model Assessment of Beta-cell Function (HOMA-B) at Year 3
Description: HOMA-B at Year 3. HOMA-B is an index of beta-cell function and was calculated as: HOMA-B = (20 x fasting insulin (measured in pmol/L))/((fasting glucose (measured in mmol/L) - 3.5) x 7.175).
Time Frame: Year 3 in Period II
Population: ITT Efficacy Population. The analysis included only time points up to that week where at least 25% of the originally enrolled population was still in the study. Missing data at Year 3 was not imputed.
Measure: Least Squares Mean (Standard Error); unit: ratio
Arm/Group | Exen + Met | Glim + Met
Number analyzed (Participants) | 148 | 166
ratio | 66.86 (4.045) | 68.52 (3.813)
Statistical Analysis 1: Comparison: Exen + Met vs Glim + Met; Mixed-model Repeated Measures (MMRM) analysis includes treatment, visit, and treatment by visit interaction, and baseline value as a covariate. The unstructured covariance matrix was used; Test type: Superiority or Other; p = 0.7648, Mixed Models Analysis; Least Squares Mean Difference = -1.66, 95% CI 2-sided [-12.58 to 9.25], Standard Error of Mean 5.560

4. Secondary Outcome: Change in HOMA-B From Baseline to Endpoint
Description: Change in HOMA-B from baseline to endpoint.
Time Frame: Baseline, end of Period II (up to 4.5 years)
Population: ITT Efficacy Population. Missing data at endpoint was imputed using last observation carried forward (LOCF) approach.
Measure: Least Squares Mean (Standard Error); unit: ratio
Arm/Group | Exen + Met | Glim + Met
Number analyzed (Participants) | 326 | 329
ratio | 5.56 (6.147) | 19.92 (6.340)
Statistical Analysis 1: Comparison: Exen + Met vs Glim + Met; Change in HOMA-B from baseline to endpoint was analyzed by an analysis of covariance (ANCOVA) model that includes treatment and baseline HbA1c stratum (<=7.3%, >7.3% to <=8.2%, >8.2%) as factors and baseline value as a covariate; Test type: Superiority or Other; p = 0.0528, ANCOVA; Least Squares Mean Difference = -14.35, 95% CI 2-sided [-28.88 to 0.17], Standard Error of Mean 7.399

5. Secondary Outcome: Fasting Proinsulin/Insulin Ratio at Year 3
Description: Fasting proinsulin (measured in pmol/L)/insulin (measured in pmol/L) ratio at Year 3.
Time Frame: Year 3 in Period II
Population: as for outcome 3
Measure: Least Squares Mean (Standard Error); unit: ratio
Arm/Group | Exen + Met | Glim + Met
Number analyzed (Participants) | 152 | 170
ratio | 0.22 (0.023) | 0.23 (0.022)
Statistical Analysis 1: Comparison: Exen + Met vs Glim + Met; MMRM analysis includes treatment, visit, and treatment by visit interaction, and baseline value as a covariate. The unstructured covariance matrix was used; Test type: Superiority or Other; p = 0.9040, Mixed Models Analysis; Least Squares Mean Difference = -0.00, 95% CI 2-sided [-0.07 to 0.06], Standard Error of Mean 0.032

6. Secondary Outcome: Change in Fasting Proinsulin/Insulin Ratio From Baseline to Endpoint.
Description: Change in fasting proinsulin (measured in pmol/L)/insulin (measured in pmol/L) ratio from baseline to endpoint.
Time Frame: Baseline, end of Period II (up to 4.5 years)
Population: ITT Efficacy Population. Missing data at endpoint was imputed using LOCF approach.
Measure: Least Squares Mean (Standard Error); unit: ratio
Arm/Group | Exen + Met | Glim + Met
Number analyzed (Participants) | 326 | 331
ratio | 0.03 (0.014) | 0.05 (0.015)
Statistical Analysis 1: Comparison: Exen + Met vs Glim + Met; Change in fasting proinsulin/insulin ratio from baseline to endpoint was analyzed by an ANCOVA model that includes treatment and baseline HbA1c stratum (<=7.3%, >7.3% to <=8.2%, >8.2%) as factors and baseline value as a covariate; Test type: Superiority or Other; p = 0.2500, ANCOVA; Least Squares Mean Difference = -0.02, 95% CI 2-sided [-0.05 to 0.01], Standard Error of Mean 0.017

7. Secondary Outcome: Ratio of the 30 Minute Increment in Plasma Insulin Concentration and the 30 Minute Increment in Plasma Glucose During the Oral Glucose Tolerance Test (DI30/DG30 Ratio) at Year 3
Description: DI30/DG30 at Year 3. DI30/DG30 ratio was calculated as (30 minute post prandial insulin - fasting insulin) (measured in pmol/L)/(30 minute post prandial glucose - fasting glucose) (measured in mmol/L).
Time Frame: Year 3 in Period II
Population: as for outcome 3
Measure: Least Squares Mean (Standard Error); unit: ratio
Arm/Group | Exen + Met | Glim + Met
Number analyzed (Participants) | 130 | 156
ratio | 25.81 (3.323) | 26.38 (3.032)
Statistical Analysis 1: Comparison: Exen + Met vs Glim + Met; [analysis description as in outcome 5, analysis 1]; Test type: Superiority or Other; p = 0.9001, Mixed Models Analysis; Least Squares Mean Difference = -0.56, 95% CI 2-sided [-9.40 to 8.27], Standard Error of Mean 4.497

8. Secondary Outcome: Change in DI30/DG30 Ratio From Baseline to Endpoint
Description: Change in DI30/DG30 ratio from baseline to endpoint.
Time Frame: Baseline, end of Period II (up to 4.5 years)
Population: ITT Efficacy Population. Missing data at endpoint was imputed using LOCF approach.
Measure: Least Squares Mean (Standard Error); unit: ratio
Arm/Group | Exen + Met | Glim + Met
Number analyzed (Participants) | 302 | 311
ratio | 12.10 (4.115) | 0.91 (4.299)
Statistical Analysis 1: Comparison: Exen + Met vs Glim + Met; Change in DI30/DG30 ratio from baseline to endpoint was analyzed by an ANCOVA model that includes treatment and baseline HbA1c stratum (<=7.3%, >7.3% to <=8.2%, >8.2%) as factors and baseline value as a covariate; Test type: Superiority or Other; p = 0.0246, ANCOVA; Least Squares Mean Difference = 11.19, 95% CI 2-sided [1.44 to 20.95], Standard Error of Mean 4.966

9. Secondary Outcome: Disposition Index at Year 3
Description: Disposition Index at Year 3. Disposition index was calculated as (DI30/DG30 ratio)/(HOMA index for insulin resistance (HOMA-IR)); where HOMA-IR=(fasting insulin (measured in pmol/L) x fasting glucose (measured in mmol/L))/(22.5 x 7.175).
Time Frame: Year 3 in Period II
Population: as for outcome 3
Measure: Least Squares Mean (Standard Error); unit: ratio
Arm/Group | Exen + Met | Glim + Met
Number analyzed (Participants) | 130 | 156
ratio | 12.56 (1.179) | 7.89 (1.078)
Statistical Analysis 1: Comparison: Exen + Met vs Glim + Met; [analysis description as in outcome 5, analysis 1]; Test type: Superiority or Other; p = 0.0036, Mixed Models Analysis; Least Squares Mean Difference = 4.67, 95% CI 2-sided [1.53 to 7.81], Standard Error of Mean 1.598

10. Secondary Outcome: Change in Disposition Index From Baseline to Endpoint
Description: Change in disposition index from baseline to endpoint.
Time Frame: Baseline, end of Period II (up to 4.5 years)
Population: ITT Efficacy Population. Missing data at endpoint was imputed using LOCF approach.
Measure: Least Squares Mean (Standard Error); unit: ratio
Arm/Group | Exen + Met | Glim + Met
Number analyzed (Participants) | 302 | 311
ratio | 9.15 (1.764) | 1.82 (1.849)
Statistical Analysis 1: Comparison: Exen + Met vs Glim + Met; Change in disposition index from baseline to endpoint was analyzed by an ANCOVA model that includes treatment and baseline HbA1c stratum (<=7.3%, >7.3% to <=8.2%, >8.2%) as factors and baseline value as a covariate; Test type: Superiority or Other; p = 0.0006, ANCOVA; Least Squares Mean Difference = 7.33, 95% CI 2-sided [3.15 to 11.50], Standard Error of Mean 2.128

11. Secondary Outcome: Change in HbA1c From Baseline to Year 3
Description: Change in HbA1c from baseline to Year 3.
Time Frame: Baseline, Year 3 in Period II
Population: as for outcome 3
Measure: Least Squares Mean (Standard Error); unit: percentage of total hemoglobin
Arm/Group | Exen + Met | Glim + Met
Number analyzed (Participants) | 182 | 197
percentage of total hemoglobin | -0.30 (0.051) | -0.12 (0.049)
Statistical Analysis 1: Comparison: Exen + Met vs Glim + Met; [analysis description as in outcome 5, analysis 1]; Test type: Superiority or Other; p = 0.0128, Mixed Models Analysis; Least Squares Mean Difference = -0.18, 95% CI 2-sided [-0.31 to -0.04], Standard Error of Mean 0.070

12. Secondary Outcome: Change in HbA1c From Baseline to Endpoint
Description: Change in HbA1c from baseline to endpoint. Endpoint for HbA1c was defined as the HbA1c measured at the treatment failure for patients reaching primary endpoint and was the last observation in study period II for other patients (either followed until the end of the study period II or discontinuing the study).
Time Frame: Baseline, end of Period II (up to 4.5 years)
Population: ITT Efficacy Population.
Measure: Least Squares Mean (Standard Error); unit: percentage of total hemoglobin
Arm/Group | Exen + Met | Glim + Met
Number analyzed (Participants) | 488 | 485
percentage of total hemoglobin | -0.36 (0.035) | -0.21 (0.035)
Statistical Analysis 1: Comparison: Exen + Met vs Glim + Met; Change in HbA1c from baseline to endpoint was analyzed by an ANCOVA model that includes treatment as factor and baseline value as a covariate; Test type: Superiority or Other; p = 0.0015, ANCOVA; Least Squares Mean Difference = -0.16, 95% CI 2-sided [-0.26 to -0.06], Standard Error of Mean 0.050

13. Secondary Outcome: Fasting Plasma Glucose at Year 3
Description: Fasting plasma glucose at Year 3.
Time Frame: Year 3 in Period II
Population: as for outcome 3
Measure: Least Squares Mean (Standard Error); unit: mmol/L
Arm/Group | Exen + Met | Glim + Met
Number analyzed (Participants) | 149 | 166
mmol/L | 7.27 (0.127) | 7.96 (0.120)
Statistical Analysis 1: Comparison: Exen + Met vs Glim + Met; MMRM includes treatment, visit, and treatment by visit interaction, and baseline value as a covariate. The unstructured covariance matrix was used; Test type: Superiority or Other; p < .0001, Mixed Models Analysis; Least Squares Mean Difference = -0.69, 95% CI 2-sided [-1.03 to -0.34], Standard Error of Mean 0.174

14. Secondary Outcome: Change in Fasting Plasma Glucose From Baseline to Endpoint
Description: Change in fasting plasma glucose from baseline to endpoint.
Time Frame: Baseline, end of Period II (up to 4.5 years)
Population: ITT Efficacy Population. Missing data at endpoint was imputed using LOCF approach.
Measure: Least Squares Mean (Standard Error); unit: mmol/L
Arm/Group | Exen + Met | Glim + Met
Number analyzed (Participants) | 327 | 329
mmol/L | -0.87 (0.155) | -0.41 (0.161)
Statistical Analysis 1: Comparison: Exen + Met vs Glim + Met; Change in fasting plasma glucose from baseline to endpoint was analyzed by an ANCOVA model that includes treatment and baseline HbA1c stratum (<=7.3%, >7.3% to <=8.2%, >8.2%) as factors and baseline value as a covariate; Test type: Superiority or Other; p = 0.0109, ANCOVA; Least Squares Mean Difference = -0.47, 95% CI 2-sided [-0.83 to -0.11], Standard Error of Mean 0.183

15. Secondary Outcome: Postprandial (2 Hours) Plasma Glucose at Year 3
Description: Postprandial (2 hours) plasma glucose at Year 3.
Time Frame: Year 3 in Period II
Population: as for outcome 3
Measure: Least Squares Mean (Standard Error); unit: mmol/L
Arm/Group | Exen + Met | Glim + Met
Number analyzed (Participants) | 138 | 160
mmol/L | 12.65 (0.311) | 15.45 (0.289)
Statistical Analysis 1: Comparison: Exen + Met vs Glim + Met; [analysis description as in outcome 5, analysis 1]; Test type: Superiority or Other; p < .0001, Mixed Models Analysis; Least Squares Mean Difference = -2.80, 95% CI 2-sided [-3.64 to -1.97], Standard Error of Mean 0.424

16. Secondary Outcome: Change in Postprandial (2 Hours) Plasma Glucose From Baseline to Endpoint
Description: Change from baseline in postprandial (2 hours) plasma glucose to endpoint.
Time Frame: Baseline, end of Period II (up to 4.5 years)
Population: ITT Efficacy Population. Missing data at endpoint was imputed using LOCF approach.
Measure: Least Squares Mean (Standard Error); unit: mmol/L
Arm/Group | Exen + Met | Glim + Met
Number analyzed (Participants) | 310 | 320
mmol/L | -2.72 (0.275) | -0.53 (0.286)
Statistical Analysis 1: Comparison: Exen + Met vs Glim + Met; Change in postprandial (2 hours) plasma glucose from baseline to endpoint was analyzed by an ANCOVA model that includes treatment and baseline HbA1c stratum (<=7.3%, >7.3% to <=8.2%, >8.2%) as factors and baseline value as a covariate; Test type: Superiority or Other; p < .0001, ANCOVA; Least Squares Mean Difference = -2.19, 95% CI 2-sided [-2.84 to -1.55], Standard Error of Mean 0.327

17. Secondary Outcome: Change in Body Weight From Baseline to Year 3
Description: Change in Body weight from baseline to Year 3.
Time Frame: Baseline, Year 3 in Period II
Population: ITT Safety Population: Enrolled patients receiving at least one dose of study medication in Study Period II with patients analyzed according to treatment actually received. The analysis included only time points up to that week where at least 25% of the originally enrolled population was still in the study. Missing data at Year 3 was not imputed.
Measure: Least Squares Mean (Standard Error); unit: kg
Arm/Group | Exen + Met | Glim + Met
Number analyzed (Participants) | 185 | 201
kg | -3.92 (0.335) | 1.47 (0.319)
Statistical Analysis 1: Comparison: Exen + Met vs Glim + Met; MMRM analysis includes treatment, visit, and treatment by visit interaction and baseline value as a covariate. The unstructured covariance matrix was used; Test type: Superiority or Other; p < .0001, Mixed Models Analysis; Least Squares Mean Difference = -5.40, 95% CI 2-sided [-6.31 to -4.49], Standard Error of Mean 0.463

18. Secondary Outcome: Systolic Blood Pressure at Year 3
Description: Systolic Blood pressure at Year 3.
Time Frame: Year 3 in Period II
Population: ITT Safety Population. The analysis included only time points up to that week where at least 25% of the originally enrolled population was still in the study. Missing data at Year 3 was not imputed.
Measure: Least Squares Mean (Standard Error); unit: mmHg
Arm/Group | Exen + Met | Glim + Met
Number analyzed (Participants) | 183 | 203
mmHg | 130.58 (0.891) | 135.78 (0.845)
Statistical Analysis 1: Comparison: Exen + Met vs Glim + Met; [analysis description as in outcome 5, analysis 1]; Test type: Superiority or Other; p < .0001, Mixed Models Analysis; Least Squares Mean Difference = -5.20, 95% CI 2-sided [-7.61 to -2.79], Standard Error of Mean 1.228

19. Secondary Outcome: Diastolic Blood Pressure at Year 3
Description: Diastolic Blood pressure at Year 3.
Time Frame: Year 3 in Period II
Population: as for outcome 18
Measure: Least Squares Mean (Standard Error); unit: mmHg
Arm/Group | Exen + Met | Glim + Met
Number analyzed (Participants) | 183 | 203
mmHg | 77.45 (0.544) | 79.16 (0.517)
Statistical Analysis 1: Comparison: Exen + Met vs Glim + Met; [analysis description as in outcome 5, analysis 1]; Test type: Superiority or Other; p = 0.0228, Mixed Models Analysis; Least Squares Mean Difference = -1.71, 95% CI 2-sided [-3.18 to -0.24], Standard Error of Mean 0.750

20. Secondary Outcome: Heart Rate at Year 3
Description: Heart rate at Year 3.
Time Frame: Year 3 in Period II
Population: as for outcome 18
Measure: Least Squares Mean (Standard Error); unit: beats per minute
Arm/Group | Exen + Met | Glim + Met
Number analyzed (Participants) | 181 | 199
beats per minute | 73.51 (0.583) | 74.23 (0.555)
Statistical Analysis 1: Comparison: Exen + Met vs Glim + Met; MMRM analysis includes treatment, visit, and visit by treatment interaction, and baseline value as a covariate. The unstructured covariance matrix was used; Test type: Superiority or Other; p = 0.3737, Mixed Models Analysis; Least Squares Mean Difference = -0.72, 95% CI 2-sided [-2.30 to 0.86], Standard Error of Mean 0.805

21. Secondary Outcome: Triglycerides at Year 3
Description: Triglycerides at Year 3.
Time Frame: Year 3 in Period II
Population: as for outcome 18
Measure: Least Squares Mean (Standard Error); unit: mmol/L
Arm/Group | Exen + Met | Glim + Met
Number analyzed (Participants) | 178 | 193
mmol/L | 1.69 (0.065) | 1.95 (0.062)
Statistical Analysis 1: Comparison: Exen + Met vs Glim + Met; [analysis description as in outcome 5, analysis 1]; Test type: Superiority or Other; p = 0.0042, Mixed Models Analysis; Least Squares Mean Difference = -0.26, 95% CI 2-sided [-0.43 to -0.08], Standard Error of Mean 0.089

22. Secondary Outcome: Total Cholesterol at Year 3
Description: Total Cholesterol at Year 3.
Time Frame: Year 3 in Period II
Population: as for outcome 18
Measure: Least Squares Mean (Standard Error); unit: mmol/L
Arm/Group | Exen + Met | Glim + Met
Number analyzed (Participants) | 178 | 193
mmol/L | 4.77 (0.057) | 4.75 (0.054)
Statistical Analysis 1: Comparison: Exen + Met vs Glim + Met; [analysis description as in outcome 5, analysis 1]; Test type: Superiority or Other; p = 0.7914, Mixed Models Analysis; Least Squares Mean Difference = 0.02, 95% CI 2-sided [-0.13 to 0.18], Standard Error of Mean 0.079

23. Secondary Outcome: High-density Lipoprotein (HDL) Cholesterol at Year 3
Description: HDL Cholesterol at Year 3.
Time Frame: Year 3 in Period II
Population: as for outcome 18
Measure: Least Squares Mean (Standard Error); unit: mmol/L
Arm/Group | Exen + Met | Glim + Met
Number analyzed (Participants) | 178 | 195
mmol/L | 1.31 (0.013) | 1.25 (0.013)
Statistical Analysis 1: Comparison: Exen + Met vs Glim + Met; [analysis description as in outcome 5, analysis 1]; Test type: Superiority or Other; p = 0.0011, Mixed Models Analysis; Least Squares Mean Difference = 0.06, 95% CI 2-sided [0.02 to 0.10], Standard Error of Mean 0.019

24. Secondary Outcome: Hypoglycemia Rate Per Year
Description: All hypoglycemia episodes were taken into account. Severe hypoglycemia: event requiring assistance of another person to administer carbohydrate, glucagons, or other resuscitative actions; Documented symptomatic hypoglycemia: event with typical symptoms accompanied by a measured plasma glucose concentration <=70 mg/dL; Asymptomatic hypoglycemia: event not accompanied by typical symptoms but with a measured plasma glucose concentration <=70 mg/dL; Probable symptomatic hypoglycemia: event with symptoms not accompanied by a plasma glucose determination.
Time Frame: Baseline to end of Period II (up to 4.5 years)
Population: ITT Safety Population.
Measure: Least Squares Mean (Standard Error); unit: events per subject-year
Arm/Group | Exen + Met | Glim + Met
Number analyzed (Participants) | 511 | 508
events per subject-year | 1.52 (0.142) | 5.32 (0.473)
Statistical Analysis 1: Comparison: Exen + Met vs Glim + Met; The number of hypoglycemic episodes by patient were compared between treatment groups using a negative binomial model with effects for treatment and baseline HbA1c and the logarithm of the days of exposure as the offset variable; Test type: Superiority or Other; p < .0001, Negative Binomial Model; Least Squares Mean Difference = 0.29, 95% CI 2-sided [0.22 to 0.37], Standard Error of Mean 0.037

25. Secondary Outcome: Change in HbA1c From Baseline to Year 2 for Patients Randomized at Entry in Period III
Description: Change in HbA1c from baseline to Year 2.
Time Frame: Baseline in Period III, Year 2 in Period III
Population: Extension ITT Efficacy Population: Extension enrolled patients with at least one post-baseline measurement of HbA1c in Study Period III. The analysis included patients randomized at entry in study period III. Missing data at Year 2 was not imputed.
Measure: Least Squares Mean (Standard Error); unit: percentage of total hemoglobin
Groups:
- Exen + Met + Glim - Randomized: Glimepiride once daily, started at 1 mg dose and titrated up to maintenance doses, was added to Exenatide 10 mcg twice daily subcutaneously injected and daily oral Metformin in Period III
- Exen + Met + Pio or Rosi - Randomized: Oral Rosiglitazone or Pioglitazone once or twice daily, started 15 mg per day, was added to Exenatide 10 mcg twice daily subcutaneously injected and daily oral Metformin in Period III
Arm/Group | Exen + Met + Glim - Randomized | Exen + Met + Pio or Rosi - Randomized
Number analyzed (Participants) | 44 | 42
percentage of total hemoglobin | -0.19 (0.099) | -0.47 (0.100)
Statistical Analysis 1: Comparison: Exen + Met + Glim - Randomized vs Exen + Met + Pio or Rosi - Randomized; MMRM analysis includes treatment, visit, and treatment by visit interaction, and baseline value at Period III as a covariate. The compound symmetric covariance structure was assumed; Test type: Superiority or Other; p = 0.0508, Mixed Models Analysis; Least Squares Mean Difference = 0.28, 95% CI 2-sided [-0.00 to 0.55], Standard Error of Mean 0.141

26. Secondary Outcome: Change in HbA1c From Baseline to Year 2 for Patients Not Randomized at Entry in Period III
Description: Change in HbA1c from baseline to Year 2.
Time Frame: Baseline in Period III, Year 2 in Period III
Population: Extension ITT Efficacy population. The analysis included patients not randomized at entry in study period III. Missing data at Year 2 was not imputed.
Measure: Mean (Standard Deviation); unit: percentage of total hemoglobin
Groups:
- Glim + Met + Exen - Not Randomized: Exenatide 10 mcg twice daily subcutaneously injected (5 mcg exenatide per dose for the first 4 weeks followed by 10 mcg exenatide per dose for the remainder of period III) was added to oral Glimepiride once daily and daily oral Metformin in Period III
Arm/Group | Glim + Met + Exen - Not Randomized
Number analyzed (Participants) | 89
percentage of total hemoglobin | -0.47 (0.984)

27. Secondary Outcome: Hypoglycemia Rate Per Year in Period III
Description: as for outcome 24
Time Frame: Start of Period III to end of study
Population: Extension ITT Safety Population: Extension enrolled patients receiving at least one dose of study medication in Study Period III.
Measure: Mean (Standard Deviation); unit: events per subject-year
Groups:
- Exen + Metformin + Glim - Randomized: Glimepiride once daily, started at 1 mg dose and titrated up to maintenance doses, was added to Exenatide 10 mcg twice daily subcutaneously injected and daily oral Metformin in Period III
Arm/Group | Exen + Metformin + Glim - Randomized | Exen + Met + Pio or Rosi - Randomized | Glim + Met + Exen - Not Randomized
Number analyzed (Participants) | 74 | 76 | 166
events per subject-year | 2.78 (5.456) | 0.60 (1.674) | 4.62 (10.411)

ADVERSE EVENTS:
Arm/Group | Period II, Glim + Met | Period III, Exen + Met + Glim - Randomized | Period III, Exen + Met + Pio or Rosi - Randomized | Period III, Glim + Met + Exen - Not Randomized | Period II, Exen + Met
Serious Adverse Events (participants affected / at risk) | 68/508 | 7/74 | 13/76 | 19/166 | 73/511
Other Adverse Events (participants affected / at risk) | 248/508 | 39/74 | 39/76 | 91/166 | 311/511
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Period II, Glim + Met (N=508) | Period III, Exen + Met + Glim - Randomized (N=74) | Period III, Exen + Met + Pio or Rosi - Randomized (N=76) | Period III, Glim + Met + Exen - Not Randomized (N=166) | Period II, Exen + Met (N=511)
Breast cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 1 | 1 | 3
Fall (Injury, poisoning and procedural complications) | 2 | 0 | 0 | 1 | 3
Nephrolithiasis (Renal and urinary disorders) | 1 | 0 | 0 | 0 | 3
Atrial fibrillation (Cardiac disorders) | 2 | 0 | 0 | 0 | 2
Cerebrovascular accident (Nervous system disorders) | 0 | 0 | 0 | 0 | 2
Cholelithiasis (Hepatobiliary disorders) | 0 | 0 | 0 | 1 | 2
Erysipelas (Infections and infestations) | 0 | 0 | 0 | 0 | 2
Ischaemic cardiomyopathy (Cardiac disorders) | 0 | 0 | 0 | 0 | 2
Lower limb fracture (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 2
Osteoarthritis (Musculoskeletal and connective tissue disorders) | 4 | 0 | 0 | 0 | 2
Prostate cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0 | 0 | 2
Renal colic (Renal and urinary disorders) | 0 | 0 | 0 | 0 | 2
Sleep apnoea syndrome (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 2
Spinal column stenosis (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0 | 0 | 2
Syncope (Nervous system disorders) | 0 | 0 | 0 | 0 | 2
Tachyarrhythmia (Cardiac disorders) | 0 | 0 | 0 | 0 | 2
Abdominal pain (Gastrointestinal disorders) | 0 | 0 | 1 | 0 | 1
Abscess (Infections and infestations) | 0 | 0 | 0 | 0 | 1
Abscess limb (Infections and infestations) | 0 | 0 | 0 | 0 | 1
Acute coronary syndrome (Cardiac disorders) | 1 | 0 | 0 | 1 | 1
Anaemia (Blood and lymphatic system disorders) | 0 | 0 | 0 | 0 | 1
Anal fissure (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 1
Angina pectoris (Cardiac disorders) | 0 | 0 | 0 | 0 | 1
Atrial flutter (Cardiac disorders) | 0 | 0 | 0 | 0 | 1
Basal cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0 | 1 | 1
Brain contusion (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 1
Bullous lung disease (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 1
Cardiac failure (Cardiac disorders) | 0 | 0 | 0 | 0 | 1
Carotid arteriosclerosis (Nervous system disorders) | 0 | 0 | 0 | 0 | 1
Cellulitis (Infections and infestations) | 0 | 0 | 0 | 0 | 1
Cervical spinal stenosis (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 1
Chest pain (General disorders) | 0 | 0 | 1 | 0 | 1
Cholecystitis (Hepatobiliary disorders) | 1 | 0 | 0 | 0 | 1
Chronic obstructive pulmonary disease (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0 | 0 | 1
Colon cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 | 0 | 0 | 1 | 1
Colonic polyp (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 1
Colorectal cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 0 | 1
Constipation (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 1
Contusion (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 1
Cystitis haemorrhagic (Renal and urinary disorders) | 0 | 0 | 0 | 0 | 1
Deep vein thrombosis (Vascular disorders) | 0 | 0 | 0 | 0 | 1
Encephalitis (Nervous system disorders) | 0 | 0 | 0 | 0 | 1
Faecaloma (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 1
Femoral neck fracture (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 1
Gallbladder cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 0 | 1
Gastroenteritis norovirus (Infections and infestations) | 0 | 0 | 0 | 0 | 1
Glioblastoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 0 | 1
HIV infection (Infections and infestations) | 0 | 0 | 0 | 0 | 1
Haemophilia A with anti factor VIII (Congenital, familial and genetic disorders) | 0 | 0 | 0 | 0 | 1
Helicobacter gastritis (Infections and infestations) | 0 | 0 | 0 | 0 | 1
Influenza (Infections and infestations) | 0 | 0 | 0 | 0 | 1
Inguinal hernia (Gastrointestinal disorders) | 1 | 0 | 0 | 0 | 1
Injury (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 1
Intervertebral disc degeneration (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 1
Ischaemic stroke (Nervous system disorders) | 0 | 0 | 0 | 0 | 1
Limb crushing injury (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 1
Lung squamous cell carcinoma stage unspecified (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 0 | 1
Myocardial infarction (Cardiac disorders) | 2 | 0 | 0 | 0 | 1
Pain in extremity (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 1
Palpitations (Cardiac disorders) | 0 | 0 | 0 | 0 | 1
Periarthritis (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1 | 1 | 1
Pneumonia (Infections and infestations) | 1 | 0 | 0 | 0 | 1
Pubis fracture (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 1
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 2 | 0 | 0 | 0 | 1
Radiculopathy (Nervous system disorders) | 0 | 0 | 0 | 0 | 1
Radius fracture (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 1
Rectal cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 0 | 1
Renal failure acute (Renal and urinary disorders) | 1 | 0 | 0 | 0 | 1
Road traffic accident (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 1
Sciatica (Nervous system disorders) | 1 | 0 | 0 | 0 | 1
Sinusitis (Infections and infestations) | 0 | 0 | 0 | 0 | 1
Sternal fracture (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 1
Subdural haemorrhage (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 1
Sudden cardiac death (General disorders) | 0 | 0 | 0 | 0 | 1
Tendon rupture (Injury, poisoning and procedural complications) | 3 | 0 | 0 | 0 | 1
Transient ischaemic attack (Nervous system disorders) | 0 | 0 | 0 | 0 | 1
Umbilical hernia (Gastrointestinal disorders) | 1 | 0 | 0 | 0 | 1
Uterine cervical erosion (Reproductive system and breast disorders) | 0 | 0 | 0 | 0 | 1
Uterine leiomyoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0 | 0 | 1
Viral labyrinthitis (Infections and infestations) | 0 | 0 | 0 | 0 | 1
Abdominal adhesions (Gastrointestinal disorders) | 1 | 0 | 0 | 0 | 0
Abdominal hernia (Gastrointestinal disorders) | 1 | 0 | 0 | 0 | 0
Accident (Injury, poisoning and procedural complications) | 1 | 0 | 0 | 0 | 0
Acute abdomen (Gastrointestinal disorders) | 1 | 0 | 0 | 0 | 0
Acute myocardial infarction (Cardiac disorders) | 2 | 0 | 0 | 0 | 0
Anal abscess (Infections and infestations) | 0 | 0 | 1 | 0 | 0
Angina unstable (Cardiac disorders) | 0 | 0 | 1 | 2 | 0
Angle closure glaucoma (Eye disorders) | 1 | 0 | 0 | 0 | 0
Appendicitis (Infections and infestations) | 1 | 0 | 0 | 0 | 0
Arthralgia (Musculoskeletal and connective tissue disorders) | 2 | 0 | 0 | 0 | 0
Asthma (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 1 | 0
Bladder cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 | 0 | 0 | 0 | 0
Bladder neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0 | 0 | 0
Breast cancer metastatic (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0 | 0 | 0
Bronchitis (Infections and infestations) | 1 | 0 | 0 | 0 | 0
Bursitis (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1 | 0 | 0
Calculus ureteric (Renal and urinary disorders) | 0 | 1 | 0 | 0 | 0
Cardiac disorder (Cardiac disorders) | 1 | 0 | 0 | 0 | 0
Carpal tunnel syndrome (Nervous system disorders) | 1 | 0 | 0 | 0 | 0
Chondropathy (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0 | 0 | 0
Clavicle fracture (Injury, poisoning and procedural complications) | 1 | 0 | 0 | 0 | 0
Coronary artery disease (Cardiac disorders) | 3 | 1 | 0 | 1 | 0
Depression (Psychiatric disorders) | 1 | 0 | 0 | 0 | 0
Dermoid cyst (Congenital, familial and genetic disorders) | 1 | 0 | 0 | 0 | 0
Diverticulum intestinal (Gastrointestinal disorders) | 1 | 0 | 0 | 0 | 0
Dyspepsia (Gastrointestinal disorders) | 1 | 0 | 0 | 0 | 0
Endometrial cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0 | 0 | 0
Endometrial hyperplasia (Reproductive system and breast disorders) | 0 | 0 | 1 | 0 | 0
Endometrial hypertrophy (Reproductive system and breast disorders) | 1 | 0 | 0 | 0 | 0
Exostosis (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1 | 0 | 0
Fibula fracture (Injury, poisoning and procedural complications) | 1 | 0 | 0 | 0 | 0
Foot deformity (Musculoskeletal and connective tissue disorders) | 1 | 0 | 1 | 0 | 0
Foot fracture (Injury, poisoning and procedural complications) | 1 | 0 | 0 | 1 | 0
Gastric neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0 | 0 | 0
Gastritis (Gastrointestinal disorders) | 0 | 0 | 0 | 1 | 0
Gastroenteritis (Infections and infestations) | 1 | 0 | 0 | 0 | 0
Gastrointestinal inflammation (Gastrointestinal disorders) | 1 | 0 | 0 | 0 | 0
Goitre (Endocrine disorders) | 3 | 0 | 0 | 0 | 0
Haemorrhoids (Gastrointestinal disorders) | 0 | 0 | 0 | 1 | 0
Hypertension (Vascular disorders) | 0 | 0 | 1 | 0 | 0
Hypoglycaemia (Metabolism and nutrition disorders) | 0 | 1 | 0 | 0 | 0
Hypokalaemia (Metabolism and nutrition disorders) | 0 | 1 | 0 | 0 | 0
Infected epidermal cyst (Infections and infestations) | 1 | 0 | 0 | 0 | 0
Intervertebral disc protrusion (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1 | 0 | 0
Intervertebral discitis (Infections and infestations) | 1 | 0 | 0 | 0 | 0
Joint effusion (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0 | 0 | 0
Knee deformity (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0 | 0 | 0
Localised infection (Infections and infestations) | 1 | 0 | 0 | 0 | 0
Macular oedema (Eye disorders) | 0 | 0 | 1 | 0 | 0
Meniscus lesion (Injury, poisoning and procedural complications) | 4 | 0 | 0 | 0 | 0
Mental disorder (Psychiatric disorders) | 0 | 0 | 0 | 1 | 0
Metastases to bone (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0 | 0 | 0
Metastases to liver (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0 | 0 | 0
Metrorrhagia (Reproductive system and breast disorders) | 1 | 0 | 0 | 0 | 0
Mood altered (Psychiatric disorders) | 1 | 0 | 0 | 0 | 0
Myocardial ischaemia (Cardiac disorders) | 1 | 0 | 0 | 1 | 0
Nervous system disorder (Nervous system disorders) | 0 | 0 | 0 | 1 | 0
Nocturia (Renal and urinary disorders) | 0 | 0 | 0 | 1 | 0
Non-cardiac chest pain (General disorders) | 0 | 0 | 0 | 1 | 0
Obesity (Metabolism and nutrition disorders) | 0 | 0 | 1 | 0 | 0
Osteitis (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0 | 0 | 0
Osteomyelitis (Infections and infestations) | 1 | 0 | 0 | 0 | 0
Ovarian cyst (Reproductive system and breast disorders) | 1 | 0 | 0 | 0 | 0
Pancreatitis (Gastrointestinal disorders) | 0 | 0 | 0 | 1 | 0
Pelvic fracture (Injury, poisoning and procedural complications) | 1 | 0 | 0 | 0 | 0
Pericarditis (Cardiac disorders) | 1 | 0 | 0 | 0 | 0
Post procedural haematoma (Injury, poisoning and procedural complications) | 1 | 0 | 0 | 0 | 0
Postoperative wound infection (Infections and infestations) | 1 | 0 | 0 | 0 | 0
Rectosigmoid cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0 | 0 | 0
Renal neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 1 | 0 | 0
Skin ulcer (Skin and subcutaneous tissue disorders) | 1 | 0 | 0 | 0 | 0
Small cell lung cancer stage unspecified (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0 | 0 | 0
Sports injury (Injury, poisoning and procedural complications) | 1 | 0 | 0 | 0 | 0
Staphylococcal sepsis (Infections and infestations) | 1 | 0 | 0 | 0 | 0
Subcutaneous abscess (Infections and infestations) | 1 | 0 | 0 | 0 | 0
Transient global amnesia (Nervous system disorders) | 1 | 0 | 0 | 0 | 0
Upper limb fracture (Injury, poisoning and procedural complications) | 1 | 0 | 0 | 0 | 0
Ureteric injury (Injury, poisoning and procedural complications) | 1 | 0 | 0 | 0 | 0
Urinary bladder polyp (Renal and urinary disorders) | 1 | 0 | 0 | 0 | 0
Urinary tract inflammation (Renal and urinary disorders) | 1 | 0 | 0 | 0 | 0
Uterine cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0 | 0 | 0
Uterine polyp (Reproductive system and breast disorders) | 1 | 0 | 0 | 0 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Period II, Glim + Met (N=508) | Period III, Exen + Met + Glim - Randomized (N=74) | Period III, Exen + Met + Pio or Rosi - Randomized (N=76) | Period III, Glim + Met + Exen - Not Randomized (N=166) | Period II, Exen + Met (N=511)
Nausea (Gastrointestinal disorders) | 11 | 10 | 9 | 38 | 147
Nasopharyngitis (Infections and infestations) | 93 | 20 | 15 | 27 | 96
Diarrhoea (Gastrointestinal disorders) | 33 | 7 | 7 | 13 | 62
Headache (Nervous system disorders) | 48 | 11 | 7 | 10 | 56
Influenza (Infections and infestations) | 35 | 7 | 6 | 8 | 54
Back pain (Musculoskeletal and connective tissue disorders) | 54 | 5 | 9 | 9 | 52
Vomiting (Gastrointestinal disorders) | 12 | 4 | 1 | 13 | 44
Bronchitis (Infections and infestations) | 31 | 2 | 7 | 5 | 34
Dyspepsia (Gastrointestinal disorders) | 14 | 4 | 0 | 14 | 26
Pharyngitis (Infections and infestations) | 21 | 2 | 2 | 5 | 26
Abdominal pain upper (Gastrointestinal disorders) | 13 | 6 | 2 | 6 | 21
Arthralgia (Musculoskeletal and connective tissue disorders) | 41 | 2 | 2 | 6 | 21
Cough (Respiratory, thoracic and mediastinal disorders) | 25 | 4 | 4 | 10 | 18
Gastroenteritis (Infections and infestations) | 13 | 4 | 3 | 9 | 18
Pain in extremity (Musculoskeletal and connective tissue disorders) | 22 | 3 | 2 | 10 | 16
Hypertension (Vascular disorders) | 24 | 6 | 3 | 9 | 15
Cystitis (Infections and infestations) | 19 | 5 | 3 | 4 | 14
Abdominal pain (Gastrointestinal disorders) | 10 | 4 | 1 | 4 | 11
Oedema peripheral (General disorders) | 11 | 0 | 5 | 2 | 6

LIMITATIONS AND CAVEATS:
Only patients who reached primary endpoint 12 months or more before the projected end of the study could enter period III.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of more than 60 days